CLINICAL TRIAL: NCT04774913
Title: Invest-CTO: Effectiveness and Safety of a Planned Investment Procedure in High-Risk CTO PCI
Brief Title: Invest-CTO PCI Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 195282
Record Dates: First submitted 2021-02-17; First posted 2021-03-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Angina Pectoris; Quality of Life; PROM
Keywords: Percutaneous coronary intervention
MeSH Terms: conditions — Angina Pectoris | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, international, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Invest CTO PCI (Experimental): A pre-planned two staged procedure in high-risk CTO PCI
  Interventions: Procedure: Chronic total occlusion(CTO) percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: Chronic total occlusion(CTO) percutaneous coronary intervention (PCI) — CTO PCI completed as a two step procedure with an initial planned CTO modification and a completion procedure after 8-12 weeks

SUMMARY:
Following unsuccessful CTO crossing a CTO modification procedure is sometimes performed. CTO PCI registries where plaque modification has been performed in some patients, report this to be safe, and associated with higher success rates at subsequent attempts.

It has never been investigated whether a planned investment procedure, with an intention that both the initial and staged completion PCI are of shorter duration, could improve safety and efficacy.

The investigators hypothesize that

1. A planned investment procedure in the treatment of CTOs will be associated with improved patient safety
2. A planned investment procedure will be associated with improved cumulative procedure success rates
3. A planned two stage procedure will be associated with improved patient experience

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Comply with the procedural and study follow-up schedule
* Planned CTO PCI in accordance with the European and American appropriateness criteria.
* CTO defined as high-risk

Exclusion Criteria:

* Non-high risk CTO
* Occlusion within a stent
* Flush aorto-ostial occlusion of RCA and Left Main (LMS)
* Limited arterial access precluding repeat procedure
* Baseline non invasive testing showing non-viable target vessel territory
* Contra-indication to dual antiplatelet therapy
* Pregnancy
* Prior radiation skin injury
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | Up to 12 weeks
  CTO PCI Procedural success, Complete technical success plus the absence of an in-hospital major adverse cardiovascular event (MACE; death, MI, or clinically driven target vessel revascularization [TVR]
Compositie safety endpoint | 30 days post procedure
  Death, myocardial infarction and procedural related complications

SECONDARY OUTCOMES:
CTO PCI technical success | At the end of staged CTO PCI completion procedure and within 3 months
  Technical success is restoration of TIMI >=2 antegrade flow with <30% residual diameter stenosis within the CTO segment
CTO PCI investment procedural success | 30 days post procedure
  Investment complete technical success
Compositie safety endpoint | 30 days post procedure
  Death, myocardial infarction and procedural related complications
Composite Clinical endpoint | 30 days, 3 & 12 months
  Cardiac death, MI , cardiovascular hospitalization and target vessel revascularization.
European Quality of Life-5 Dimensions | Baseline, 3 and 12 months
  5 item measure of mobility, self-care, usual activity, pain or discomfort, and anxiety or depression . Score 0-100, where high score better.
Seattle angina questionnaire (SAQ7) | Baseline, 3 & 12 months
  3 domain score of physical limitation (SAQ7-PL), angina frequency (SAQ7-AF) and quality of life (SAQ7-QL). Score 0-100, where high score better.
Patient related outcome measures (PROM) | Through study completion, an average of 15 months.
  Qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Margaret B Mcentegart, PhD, Principal Investigator — Golden Jubilee National Hospital; Anja Øksnes, MD, Principal Investigator — Haukeland University Hospital
Locations (5):
- Columbia University Medical Center/ NewYork Presbyterian Hospital, New York, New York, United States
- Haukeland University Hospital, Bergen, Bergen, Norway
- United Kingdom (3):
  - Golden Jubilee National Hospital, Glasgow, Glasgow
  - Bristol Health, Bristol
  - St George´s Hospital, London

IPD SHARING:
Plan to Share IPD: No